CLINICAL TRIAL: NCT05715567
Title: Re-EValuating the Inhibition of Stress Erosions (REVISE) - COVID-19 Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19 REVISE_Cohort_22
Record Dates: First submitted 2023-02-03; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; GastroIntestinal Bleeding
Keywords: COVID-19; pandemic; gastrointestinal bleeding; pneumonia; Clostridioides difficile
MeSH Terms: conditions — COVID-19; Gastrointestinal Hemorrhage; Pneumonia | interventions — Reoperation; Clinical Trials as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COVID-19
  Interventions: Other: Re-EValuating the Inhibition of Stress Erosions (REVISE) Trial (NCT03374800)
- Patients without COVID-19
  Interventions: Other: Re-EValuating the Inhibition of Stress Erosions (REVISE) Trial (NCT03374800)

INTERVENTIONS:
Other: Re-EValuating the Inhibition of Stress Erosions (REVISE) Trial (NCT03374800) — Following the intervention of the Re-EValuating the Inhibition of Stress Erosions (REVISE) Trial (NCT03374800)

SUMMARY:
Commonly employed medications used in critically ill patients requiring life support include proton pump inhibitors (PPIs). These medications are thought to prevent gastrointestinal (GI) bleeding from stress-induced ulceration. Despite their widespread use, they do hold some risks which include infection in the form of pneumonia and diarrheal illnesses such as Clostridioides difficile infection (C. difficile). Emerging high-quality studies suggest PPI usage does not influence susceptibility to COVID-19 infection, however some studies suggest PPI use leads to poor outcomes in this population, including prolonged time on life-support and death. While we can appreciate the negative effects of PPI may be magnified in the sickest of patients, namely hospitalized patients with COVID-19, the beneficial or potentially harmful role they play in this population remains unclear.

We aim to build a clinical profile to further describe critically ill patients with COVID-19 in Ontario using the infrastructure of an ongoing multicenter clinical trial of acid suppression. We will identify characteristics that predict poor outcomes among sick COVID patients, examining the impact of PPIs on this population.

DETAILED DESCRIPTION:
The overall aims are to further characterize the high-risk population of COVID-19 patients nested within the multicenter REVISE trial. Specifically, we plan 1) to explore the impact of PPIs on mechanically ventilated critically ill COVID-19 patients, 2) describe the clinical course for patients with COVID-19 and identify characteristics that predict poor prognosis, and 3) compare outcomes to patients without COVID-19. The overall research questions are as follows:

1. Do critically ill patients projected to receive mechanical ventilation for >48 hours with COVID-19 have different clinical outcomes without PPIs?
2. Are there prognostically relevant demographic, biomarker and clinical data to characterize critically ill patients with COVID-19?
3. Do critically ill patients with COVID-19 have significant higher rates of clinically important GI bleeding, 90-day mortality, and rates of infection when compared to a propensity-matched non-COVID REVISE cohort?

To accomplish this, the investigators propose to gather information in patients' medical charts including biomarkers drawn by the ICU team, venous thromboembolism (VTE) and tracheostomy timing, to link with extensive baseline characteristics and outcomes already collected in the REVISE trial (NCT03374800)

ELIGIBILITY:
Inclusion Criteria:

Adults ≥18 years old projected to receive invasive mechanical ventilation for ≥48 hours according to the treating physician

Exclusion Criteria:

1. Already received invasive mechanical ventilation >72 hours during this hospital admission
2. Acid suppression for active gastrointestinal bleeding or high risk of bleeding (e.g., current bleeding, peptic ulcer bleeding within 8 weeks, recent severe esophagitis, Barrett's esophagus, Zollinger-Ellison syndrome); [dyspepsia or gastroesophageal reflux is not an exclusion criterion]
3. Acid suppression in the intensive care unit for >1 daily dose equivalent of a proton pump inhibitor or histamine-2-receptor antagonist
4. Dual antiplatelet therapy
5. Combined antiplatelet and therapeutic anticoagulation
6. Pantoprazole contraindication per local product information
7. Palliative care or anticipated withdrawal of advanced life support
8. Pregnancy
9. Previous enrolment in REVISE, or a related trial, or trial for which co-enrolment is prohibited
10. Patient, proxy or physician declines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible according to the inclusion and exclusion criteria of the REVISE trial, regardless of COVID status
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically important gastro-intestinal bleeding | 90 days
  The primary efficacy outcome is clinically important GI bleeding occurring in the ICU or resulting in ICU readmission during the index hospital stay.
  The definition of clinically important GI bleeding is overt GI bleeding (i.e., hematemesis, frank blood or coffee ground nasogastric aspirate, melena or hematochezia) plus 1 of the following in the absence of other causes:
  1. Hemodynamic change defined as a spontaneous decrease in invasively monitored mean arterial pressure or non-invasive systolic or diastolic blood pressure of >20 mmHg, or an orthostatic increase in pulse rate of >20 beats/minute and a decrease in systolic blood pressure of >10 mmHg, with or without vasopressor initiation or increase;
  2. vasopressor initiation;
  3. hemoglobin decrease of >2 g/dl (20 g/L) within 24 h of bleeding;
  4. transfusion of >2 units red blood cells within 24 h of bleeding; or
  5. therapeutic intervention (e.g., therapeutic endoscopy, angiography, surgery).
Primary Safety Outcome: 90 Day Mortality | 90 days after randomization
  Mortality status at day 90 post randomization

SECONDARY OUTCOMES:
Ventilator-associated pneumonia | 90 Days (while in ICU,censored at 90 days after randomization)
  VAP is diagnosed in patients who received invasive mechanical ventilation for >48 hours when there is a new, progressive or persistent radiographic infiltrate plus at least 2 of the following without other obvious cause: 1) fever (temperature>38 °C) or hypothermia (temperature <36 °C); 2) leukopenia (<4.0x106/L) or leukocytosis (>12x106/L); 3) purulent sputum; or 4) gas exchange deterioration.
C. difficile infection | 90 days (during the index hospital admission, censored at 90 days)
  Defined as clinical features (diarrhea [>3 episodes of unformed stools or Bristol type 6 or 7), ileus, or toxic megacolon) and either microbiological evidence of toxin-producing C. difficile or pseudomembranous colitis on colonoscopy in hospital.
Renal replacement therapy | While in ICU,censored at 90 days after randomization
  Defined as initiation of new renal replacement therapy in the ICU.
Hospital mortality | While in hospital, censored at 90 days after randomization
  Defined as all-cause mortality in hospital.
Patient important GI bleeding | Censored at 90 days after randomization
  Defined as overt GI bleeding, plus an invasive intervention (e.g., therapeutic endoscopy, angiography, surgery), acknowledging how some clinically important GI bleeds in prior studies did not actually require any tests or treatments, and thus may not be important to patients. This outcome will be refined by an ongoing mixed methods study with an overarching instrument-building aim.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Cook, MD, Principal Investigator — McMaster University; Brittany Dennis, MD, Principal Investigator — McMaster University
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dennis BB, Thabane L, Heels-Ansdell D, Dionne JC, Binnie A, Tsang J, Guyatt G, Ahmed A, Lauzier F, Deane A, Arabi Y, Marshall J, Zytaruk N, Saunders L, Finfer S, Myburgh J, Muscedere J, English S, Ostermann M, Hardie M, Knowles S, Cook D; REVISE Investigators the Canadian Critical Care Trials Group. Proton pump inhibitors in critically ill mechanically ventilated patients with COVID-19: protocol for a substudy of the Re-EValuating the Inhibition of Stress Erosions (REVISE) Trial. Trials. 2023 Aug 30;24(1):561. doi: 10.1186/s13063-023-07589-2. PMID 37644556